CLINICAL TRIAL: NCT06064643
Title: The Lived Experience of People With Von Willebrand Disease
Acronym: VWD360
Status: Completed | Type: Observational
Sponsor: Haemnet (Other)
Collaborators: Hemab ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: v1.0 dated 15 June 2023
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Von Willebrand Diseases
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Survey Arm: All participants will be asked to complete an online survey
  Interventions: Other: Online Survey
- Interview Arm: A sample of the survey group will be asked to take part in a single qualitative interview
  Interventions: Other: Qualitative Interview
- Bleed Diary Arm: A sample of the survey group will be asked to take part in a 30 day bleed diary
  Interventions: Other: Bleed Diary

INTERVENTIONS:
Other: Online Survey — All participants will be asked to complete an online survey
  Groups: Survey Arm
Other: Qualitative Interview — 30 survey participants will take part in a single one-hour qualitative interview.
  Groups: Interview Arm
Other: Bleed Diary — 50 participants will complete a 30 day bleed diary
  Groups: Bleed Diary Arm

SUMMARY:
von Willebrand disease (vWD) is reported to be the most common bleeding disorder, with prevalence estimated at 1% of the general population. Despite this, little is known about its natural history, or of the impact it has on affected individuals and their families.

The Haemnet vWD360 programme is a mixed-methods, natural history study designed to gain a greater understanding of vWD and its impact on individuals and their families. It comprises both qualitative and quantitative approaches and is designed to include the perspectives of individuals with a diagnosis of any subtype of vWD.

The vWD360 study includes three components:

* Quantitative cross-sectional survey
* Qualitative one-to-one interviews with affected individuals
* 30-day bleed diary.

DETAILED DESCRIPTION:
von Willebrand Disease (vWD) is an inherited blood clotting (coagulation) disorder characterized by a reduction (quantitative) or poor function (qualitative) defect of factor VIII (FVIII) and/or von Willebrand factor (vWF). There are numerous subtypes categorised as:

* Type 1: a quantitative defect characterised by decreased levels of vWF in the circulation. Many affected individuals have a mild bleeding phenotype but may have heavy menstrual bleeding (HMB) and bleed following trauma/surgery.
* Type 2: a qualitative defect that is further divided into four subtypes
* Type 2A - vWF is unable to bind to form the large vWF multimers required for coagulation
* Type 2B - vWF has enhanced binding to platelet glycoprotein Ib (GPIb), causing rapid clearance of platelets and an associated thrombocytopenia
* Type 2M - vWF has a decreased ability to bind to GPIb
* Type 2N - there is a deficiency of vWF binding to FVIII
* Type 3: the most severe vWD subtype, characterised by complete absence of vWF production and an inability to bind with FVIII, resulting in a severely reduced FVIII level.

Acquired vWD can develop as an autoimmune disorder, as a result of cancer, some cardiac conditions or following of certain drugs. It will not be considered as part of this study.vWD is characterized by prolonged or spontaneous bleeding from birth. Affected individuals tend to bruise easily, may have frequent nosebleeds (epistaxis), may bleed from the gums, bleeding within tissues (haematoma), in the gastrointestinal tract (more common later in life) and joint bleeds (in Type 3). vWD causes prolonged bleeding following injury, trauma, or surgery (including dental work). Women with vWD can have prolonged heavy menstrual bleeding, they may also have an increased risk of excessive blood loss during pregnancy and childbirth.

The severity and frequency of the bleeding episodes in vWD can vary greatly among affected individuals, even within the same family. The bleeding phenotype correlates to some degree with the subtype of VWD, with those with the severest form (Type 3) having the most bleeding.

Treatment varies based on the diagnosis. In Types 1 and 2 vWD treatment is usually 'on-demand' (after bleeding occurs) with some patients receiving prophylaxis if they have significant frequent bleeding. On demand treatment may be with oral, intra-nasal or subcutaneous treatments or with intravenous infusions of clotting factor concentrates containing FVIII/vWF. This is the method of treatment for all bleeding and prophylaxis in Type 3 vWD, where for some patients, treatment may be given at home.

The lack of routine prophylaxis in Type 1 and 2 vWD means that most patients are reliant on hospital delivered care, which may involve frequent clinic appointments, causing prolonged bleeding due to a lack of timely administration of treatment. This can result in concurrent illnesses such as iron deficiency anaemia, which further impacts on the quality of life of affected individuals and their families.

There remains a need for a comprehensive understanding of the experience of people with vWD across the whole spectrum of subtypes in order to identify:

* The nature and range of symptoms that people experience and how these vary with the different disease subtypes
* The variability in pathways through which patients progress to access appropriate care
* The impact of living with vWD on the individual's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 16 and above (UK and Ireland) and adults aged over 18 (in USA) with a confirmed diagnosis of inherited vWD of known diagnostic subtype and vWF level.
* For the qualitative interview-based substudy, 30 adults who have completed the survey and who wish to be interviewed will be purposively selected for a broad range of ages and diagnostic subtype.
* For the bleed diary substudy, 50 adults who have completed the survey and who wish to take part will be purposively selected for a broad range of ages and diagnostic subtype.

Exclusion Criteria:Participants will be excluded from the study if they:

* Have acquired vWD
* Have other inherited bleeding disorders
* Do not wish to participate in or to consent to the study.

Those for whom written/spoken English would prohibit participation will also be excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with a confirmed diagnosis of von Willebrands disease, aged 16 yrs and older (18 yrs and older in the US).
Sampling Method: Non-Probability Sample
Enrollment: 611 (Actual)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Bleeding Episodes | Survey - The month prior to completing the survey. Bleed Diary - 30 days from consent.
  To identify differences in bleeding type and rate between sub-types of vWD
Pain experiences | Survey - The month prior to completion of the survey
  To identify evidence of chronic and acute pain between sub-types of vWD
Daily Activities | Survey - one month prior to completion of the survey. Interview - life historical
  To identify differences in daily activity between sub-types of vWD

CONTACTS AND LOCATIONS:
Overall Officials: Simon Fletcher, MA, Principal Investigator — Haemnet
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom